CLINICAL TRIAL: NCT02717637
Title: Gastrointestinal Uptake of Oxycodone After Caesarean Section in Spinal Anesthesia
Brief Title: Oxycodone in Serum After Postoperative Oral Oxycodone in Caesarean Sections Under Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Dahl, Professor 2, University Hospital, Akershus
Other Study IDs: 2014/1781
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Analgesic Adverse Reaction; Cesarean Delivery Affecting Newborn
Keywords: oxycodone, caesarean, spinal anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum from blood
Oversight: Data Monitoring Committee: No

SUMMARY:
All patients undergoing an elective caesarean section under spinal anesthesia will, according to the hospital routines, receive 10 mg oxycodone slow-release tablet when arriving at our postoperative care unit (PACU). Blood samples will be taken at 0 hour, 1 hour, 2 and 6 hours after administration in order to investigate bioavailability.

DETAILED DESCRIPTION:
After written informed consent, blood samples will be taken before administration, after 1 hour, 2 hours and 6 hours. Need of rescue analgesia (morphine iv) and level of pain, as well as side effects will be registered

ELIGIBILITY:
Inclusion Criteria: Healthy women > 18 years old, with one healthy fetus scheduled for a elective caesarean section in spinal anesthesia, read and signed informed consent

-

Exclusion Criteria:

* Known intolerability to oxycodone. Previous use of opioids. Hight < 150 cm, preconceptual BMI > 35. ASA > 2.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with single fetus in cephalated position admitted for elective caesarean section in spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
level of oxycodone in serum | 1 hour after administration
level of oxycodone in serum | 2 hours after administration
level of oxycodone in serum | 6 hours after administration

SECONDARY OUTCOMES:
level of pain | 0, 1, 2, and 6 hours after administration
  NRS scale 0-10

OTHER OUTCOMES:
Side effects | 1,2 and 6 hourd after administration
  nausea and vomiting, other side effects

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Dahl, PhD, Principal Investigator — Head of anesthesia dept
Locations (1):
- Akershus University Hospital, Nordbyhagen, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No